CLINICAL TRIAL: NCT06370364
Title: Contributing Factors Affecting Nurses' Practice of Safe Blood Transfusion in Surgical and Critical Care Units
Brief Title: Nurses' Practice of Safe Blood Transfusion in Surgical and Critical Care Units
Status: Completed | Type: Observational
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Other Study IDs: 25
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Practice Nurse's Scope; Blood Transfusion
Keywords: Nurses; Employment; Contributing factors; Practice; Blood; Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nurses' Practice of Safe Blood Transfusion — Nurses' Practice of Safe Blood Transfusion

SUMMARY:
Blood transfusions are an important part of nursing procedure. Nurses play a key role in safely administering blood products to patients in surgical and critical care unit

DETAILED DESCRIPTION:
The aim of the study was to evaluate nurses' employment conditions as contributing factors affecting nurses' practice of safe blood transfusion in surgical and critical care units in Alexandria Main University Hospital.

ELIGIBILITY:
Inclusion Criteria:

Nurses

* willing to participate in the study
* work in surgical and critical care units
* Sign a consent

Exclusion Criteria:

* Nurses

  * Work in outpatient units and other units
  * Did not sign a consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A convenience sampling was utilized to recruit 350 nurses from surgical and critical care units
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure factors affecting safe blood transfusion | one month
  Factors affecting safe blood transfusion as assessed using a binary scale (Yes=1 and No=0)
observational checklist to measure nurses' practice of safe blood transfusion | three months
  Nurses' practice of safe blood transfusion as assessed using scoring of the practice checklist (zero score for not done, 0.5 score for incompletely done and one score for completely done).

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Hanaa Abbass, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University , Egypt; Maysa Elbiaa, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University , Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No